CLINICAL TRIAL: NCT02404506
Title: Eribulin as 1st Line Treatment in Elderly Patients (≥ 70 Years) With Advanced Breast Cancer: a Multicenter Phase II Trial
Brief Title: Eribulin as 1st Line Treatment in Elderly Patients With Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was prematurely terminated as of 22.07.2021 as per SAKK board decision board decision from 14th of November 2020. The trial was terminated after the primary endpoint was analyzed, which was the case end of December 2020.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 25/14; 000001310 (Other: SNCTP)
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; Adenocarcinoma
Keywords: Eribulin; Breast Cancer; Elderly Patient; Phase II Trial; HER2-neg; adenocarcinoma
MeSH Terms: conditions — Breast Neoplasms; Adenocarcinoma | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm: Eribulin mesilate (Experimental)
  Interventions: Drug: Eribulin mesilate

INTERVENTIONS:
Drug: Eribulin mesilate — Eribulin mesiylate 1.1mg/m2 d1, 8 every 3 weeks until Progressive disease PD
  Other Names: Halaven

SUMMARY:
Breast cancer is the most frequent malignancy in women, world-wide the leading cause of cancer mortality. One of the strongest risk factors for developing breast cancer is age, with a prevalence approaching 7% in women >70 years; more than 40% of breast cancer patients are older than 65 years. Although the survival rate has increased in the last years, about one third of patients will relapse with distant metastases. Treatment for patients with metastatic breast cancer is palliative, therefore maintaining or improving quality of life.

The use of taxanes and anthracyclines as first line chemotherapy regimen for metastatic breast cancer is widely accepted. Both taxanes and anthracyclines have considerable side effects, especially in elderly patients.

Eribulin, a synthetic analogue of a chemotherapeutically active compound derived from the sea sponge Halichondria okadai, acts as an inhibitor of microtubule dynamics. It is registered as palliative chemotherapy in advanced breast cancer after anthracyclines and taxanes. Studies with eribulin treatment have shown similar efficacy compared to anthracyclines and taxanes, but less toxicity. Those studies showed that often the dose of eribulin had to be reduced during treatment due to toxicity without compromising the efficacy of the treatment.

The main objective of the trial is to explore the efficacy of a reduced starting dose of eribulin as first-line treatment in elderly metastatic breast cancer patients. The secondary objective of the trial is to investigate the safety of eribulin in those patients.

Eribulin mesilate 1.1mg/m2 i.v. will be administered intravenously every 3 weeks on day 1 and day 8 until progressive disease.

DETAILED DESCRIPTION:
Due to a rising number of elderly patients, fit for chemotherapy, investigating a well-tolerated and effective first line treatment is warranted. In this specific population often there are contra-indications for the use of standard first line drugs like anthracyclines and taxanes due to comorbidities (e.g. cardiac impairment or Peripheral neuropathy). Response rates in first line treatment with taxanes and anthracyclines usually do not exceed 30%. Eribulin has shown a response rate of 29% and a clinical benefit rate (corresponding to the investigators primary endpoint) of 52% in first line, so the investigators expect similar efficacy, but less toxicity.

Optimal dose, schedule and tolerability of this drug in the first line setting are unknown in the elderly population. No information on dose modifications in this population is available. Based on the data of eribulin in the first line with higher efficacy in those patients with dose reductions, the SAKK 25/14 trial investigates the reduced starting-dose of eribulin of 1.1mg/m2 for this vulnerable population of elderly patients. Growth factors to maintain a certain dose level of eribulin are not recommended, respecting the international guidelines.

SAKK has a tradition in conducting trials in the elderly population, such as SAKK 25/99 in metastatic breast cancer, SAKK 38/08 in aggressive B-cell-Lymphoma, SAKK 41/10 in metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must give written informed consent according to ICH/GCP regulations before registration
* Histologically or cytologically confirmed locally advanced or metastatic HER2-neg, hormone receptor positive or negative adenocarcinoma of the breast with measurable or evaluable disease according to RECIST 1.1 criteria
* At least 6 months since last adjuvant/neoadjuvant chemotherapy administration before registration
* At least 2 weeks since prior radiotherapy or endocrine therapy and complete recovery from these interventions at time of registration
* Baseline C-SGA and patient-reported outcome (PRO) forms have been completed
* Female patient at the age of ≥70 years
* WHO performance status 0-2
* Adequate hematological values: hemoglobin ≥80 g/L (transfusions are allowed), neutrophils ≥1.5 x 109/L, platelets ≥ 100 x 109/L
* Adequate hepatic function: bilirubin ≤1.5 x ULN, AST ≤3 x ULN, alkaline phosphatase (AP) ≤2.5 x ULN (in case of liver metastases ≤5 x ULN or in case of bone metastases ≤10 x ULN)
* Adequate renal function (calculated creatinine clearance >40 mL/min, according to the formula of Cockcroft-Gault)

Exclusion Criteria:

* Known CNS metastases
* Previous malignancy within 3 years with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
* Prior chemotherapy for advanced disease
* Concurrent anticancer treatment or treatment in a clinical trial within 30 days prior to registration. Exception: participation in SAKK 96/12
* Palliative irradiation prior to study entry with more than 30% of marrow-bearing bone irradiated
* Pre-existing neuropathy ≥G2 (according to CTCAE v4.0) at registration
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV (see Appendix 4), unstable angina pectoris, history of myocardial infarction within the last three months, significant arrhythmias, congenital long QT-syndrome)
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information
* Known hypersensitivity to trial drug or to any component of the trial drug
* Any serious underlying medical condition (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes)
* Psychiatric disorder precluding understanding of trial information, giving informed consent, taking part in the geriatric assessment, or interfering with compliance/with the trial protocol
* Any familial, sociological or geographical condition potentially hampering proper staging and compliance with the trial protocol

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Disease Control (DC) | 24 weeks
  A patient has DC, if she has complete response (CR) or partial response (PR) at any time point during treatment, or if she has stable disease (SD) for at least 24 weeks (according to RECIST v1.1).

SECONDARY OUTCOMES:
Time to treatment failure (TTF) | at treatment discontinuation (at the latest 5 years after registration)
  time from registration until treatment discontinuation due to any reason or the occurrence of a second tumor. Patients still on treatment will be censored at the date of their last eribulin administration
Objective response (OR) | at treatment discontinuation (at the latest 5 years after registration)
  A patient is defined as having OR, if she has CR or PR according to RECIST v1.1 at any time point during treatment.
  For the primary analysis, all responses (CR, PR) will be considered, including unconfirmed responses. In a sensitivity analysis, only those responses for which a confirmatory measurement at least 4 weeks later is available will be counted as CR or PR
Time to progression (TTP) | at time of progression, death or treatment discontinuation (at the latest 5 years after registration)
  TTP is defined as time from registration until documented progression according to RECIST v1.1 or death due to tumor.
  Patients not experiencing an event and patients starting a new anticancer therapy in the absence of an event will be censored at the date of their last available tumor assessment showing non-progression.
Overall survival (OS) | at time of death (at the latest 5 years after registration)
  OS is defined as time from registration until death from any cause. Patients not experiencing an event will be censored at the last date they were known to be alive.
Adverse events (AEs) | until 30 days after last dose of treatment and resolution of all related AEs thereafter (at the latest 5 years after registration)
  AEs will be assessed according to NCI CTCAE v4.0.
Patient reported neuropathy (PRO Form) and characterization of patients based on cancer-specific geriatric assessment (C-SGA) | at the first follow-up visit (at the latest 5 years after registration)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Hasler-Strub, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (26):
- Switzerland (26):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Praxis für ambulante Tumortherapie, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Klinik Engeried / Oncocare, Bern
  - Inselspital, Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Frauenfeld / Brustzentrum Thurgau, Frauenfeld
  - HFR Fribourg - Hôpital cantonal, Fribourg
  - Clinique de Genolier, Genolier
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Clinica Sant'Anna - Oncologia Varini & Calderoni & Christinat, Lugano
  - Kantonsspital Luzern, Luzerne
  - Onkologie Zentrum Spital Männedorf, Männedorf
  - Kantonsspital Olten, Olten
  - Onkologiepraxis Dr. med. Isabella Schönenberger, Sankt Gallen
  - Tumorzentrum ZeTUP, Sankt Gallen
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Rundum Onkologie am Bahnhofpark, Sargans
  - Onkologiezentrum Bürgerspital Solothurn, Solothurn
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum - Klinik im Park, Zurich
  - Brust-Zentrum AG Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No